CLINICAL TRIAL: NCT02767687
Title: Influence of Non Invasive Mechanical Ventilation on Tissue Perfusion in Patients After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Natasha de Oliveira Marcondi, Principal Investigator, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1.156.460
Record Dates: First submitted 2016-03-28; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Heart Diseases; Coronary Artery Disease
Keywords: Postoperative Care; Postoperative Period; Heart Surgery
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noninvasive ventilation (NIV) (Experimental): Noninvasive mechanical ventilation is a resource used to treat respiratory failure or to reestablish respiratory comfort and function. It is commonly used in the ICU with a regular mechanical ventilator and is offered using an interface that connects the machine to the patient. The interface used for adults and in this study, was a silicon facial mask that covers the nose and mouth of the patient, allowing him or her to open the eyes.
  Interventions: Other: Noninvasive ventilation

INTERVENTIONS:
Other: Noninvasive ventilation — Twenty minutes after extubation all subjects will receive noninvasive ventilation delivered through a facial mask with an ICU ventilator with NIV option for 60 minutes. NIV associates pressure support ventilation (PSV: 5 to 15 cmH2O) and positive end expiratory pressure (PEEP: 5 to 10 cmH2O).
  Other Names: NIV

SUMMARY:
This study evaluates whether noninvasive ventilation with continuous positive airway pressure affects tissue perfusion in patients after cardiac surgery.

DETAILED DESCRIPTION:
Patients submitted to open chest cardiac surgery will be enrolled after ICU admission. These patients will be submitted to noninvasive mechanical ventilation with continuous positive airway pressure right after extubation and tissue perfusion markers (central venous oxygen saturation (SVcO2) and lactate) will be obtained via central venous catheter.

Noninvasive mechanical ventilation is a common resource in the ICU to reduce extubation failures and to improve clinical outcomes, whether it can influence tissue perfusion remains unclear.

This study evaluates whether noninvasive ventilation affects tissue perfusion and whether tissue perfusion markers in the ICU are correlated with better clinical results for patients after heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of central venous catheter
* Invasive arterial pressure catheter
* Invasive mechanical ventilation

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Morbid obesity
* Hemodynamic instability
* Spontaneous breathing
* Need of invasive mechanical ventilation for more than 24 hours
* Intolerance to noninvasive mechanical ventilation
* Extubation failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of central venous oxygen saturation to determine tissue perfusion | Through study completion, an average of 1 year
  All patients will be admitted in ICU after surgery and will be submitted to four blood collections from the central venous catheter at different times to evaluate central venous oxygen saturation. Time 1: at ICU admission in mechanical ventilation. Time 2 : twenty minutes after extubation, before the noninvasive ventilation protocol, while breathing spontaneously with a 40% oxygen mask. Time 3: At 60 minutes of noninvasive ventilation protocol. Time 4: twenty minutes after noninvasive ventilation protocol complete while breathing spontaneously with a 40% oxygen mask. The results will be compared between then to assess if there are changes under influence of non invasive ventilation.
Evaluation of arterial lactate to determine tissue perfusion | Through study completion, an average of 1 year
  All patients will be admitted in ICU after surgery and will be submitted to four blood collections from the arterial invasive catheter at different times to evaluate arterial lactate. Time 1: at ICU admission in mechanical ventilation. Time 2 : twenty minutes after extubation, before the noninvasive ventilation protocol, while breathing spontaneously with a 40% oxygen mask. Time 3: At 60 minutes of noninvasive ventilation protocol. Time 4: twenty minutes after noninvasive ventilation protocol complete while breathing spontaneously with a 40% oxygen mask. The results will be compared between then to assess if there are changes under influence of non invasive ventilation.

SECONDARY OUTCOMES:
Respiratory complications during hospitalization | Through study completion, an average of 1 year
  Respiratory events as pleural effusion and atelectasis will be evaluated by a professional blind to the protocol of study and will be recorded.
Hemodinamycs complications during hospitalization | Through study completion, an average of 1 year
  Hemodinamycs events as arrhythmia, hypotension and cardiac arrest will be evaluated by a professional blind to the protocol of study and will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Solange Guizilini, PhD, Study Director — Federal University of São Paulo

IPD SHARING:
Plan to Share IPD: No
No participant data will be made available, however every subject was provided the investigator's e-mail address as well a phone number and was encouraged to call or send an e-mail in case of doubt or to receive information regarding the research.

REFERENCES:
- [Derived] Marcondi NO, Rocco IS, Bolzan DW, Pauletti HO, Begot I, Anjos NR, Moreira RSL, Nasrala ML, Arena R, Gomes WJ, Guizilini S. Noninvasive Ventilation After Coronary Artery Bypass Grafting in Subjects With Left-Ventricular Dysfunction. Respir Care. 2018 Jul;63(7):879-885. doi: 10.4187/respcare.05851. Epub 2018 Jun 12. PMID 29895702